CLINICAL TRIAL: NCT06114121
Title: Comparing Intrathecal Morphine and Erector Spinae Plane Regional Anesthesia Against Intrathecal Morphine Alone for Post-Cesarean Section Pain
Brief Title: Intrathecal Morphine vs. Intrathecal Morphine and Regional Anesthesia After Cesarean Section.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study will no longer be conducted
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Reine Zbeidy, Associate Professor of Clinical Anesthesiology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230857
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Post-operative Pain
Keywords: erector spinae plane block
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine; Ropivacaine; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- erector spinae plane block (Experimental): participants will be in this group for up to 9 months and receive erector spinae plane (ESP) block
  Interventions: Procedure: erector spinae plane block (ESP); Drug: Duramorph; Drug: Ropivacaine; Drug: Bupivacaine Injection
- standard of care (Experimental): participants in this group will receive the standard of care treatment and will be in this group for up to 9 months.
  Interventions: Drug: Duramorph; Drug: Ropivacaine; Drug: Bupivacaine Injection

INTERVENTIONS:
Procedure: erector spinae plane block (ESP) — nerve block for abdominal pain. administered once immediately prior to spinal anesthetic standard of care.
  Arms: erector spinae plane block
Drug: Duramorph — 100 micrograms (mcg) of morphine administered in the spinal medications one time.
Drug: Ropivacaine — Ropivacaine 0.5% between 20-40 milliliters will be administered once in the ESP block (in the spine) depending on patient weight to keep under the maximum dose.
Drug: Bupivacaine Injection — Bupivacaine 0.75% 1.4-1.7 milliliters (10-12 milligrams) spinal medication. administered one time.

SUMMARY:
The objective of the study is to optimize post-operative analgesia and improve patient satisfaction while reducing total opioid consumption after cesarean section

ELIGIBILITY:
Inclusion criteria:

* Able to consent
* BMI<35

Exclusion Criteria:

* Adults unable to consent
* BMI>35
* Individuals <18 years of age at time of admission
* Individuals taking anticoagulant medications
* Significant co-morbid disease of pregnancy (including: gestational diabetes and significant abnormal placentation)
* Pre-existing chronic pain or pain disorder diagnosis
* Conversion from neuraxial to general anesthesia
* Prisoners

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-10 (Estimated); Primary Completion 2024-09-10 (Estimated); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
post-operative opioid analgesic medication | up to 24 hours
  measurement (milligrams)

SECONDARY OUTCOMES:
change in post-operative pain medication by visual analog scale | baseline, up to 24 hours
  Patient administered instrument to indicate pain on a level from 0 to10. (0: no pain. 10: worst imaginable pain)
number of minutes to first use of rescue medication | up to 24 hours
  the number of minutes calculated using the kaplan-meier. Calculated using the number of patients that did not need the rescue analgesic at the start of each day post-surgery, and the number of patients who needed the rescue analgesic.
obstetric quality of recovery scale | up to 24 hours
  responses range from 0-10. zero is strongly agree, strongly disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Reine Zbeidy, MD, Principal Investigator — University of Miami

IPD SHARING:
Plan to Share IPD: No